CLINICAL TRIAL: NCT03230526
Title: Brain Microglial Activation in the Early Stage of the Parkinson's Disease: a Predictive Biomarker of the Evolution?
Brief Title: Identification of a Biomarker Predictive of Evolution of Parkinson Disease
Acronym: GLIAPARK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC17_0012; 2017-000411-16 (EudraCT Number)
Record Dates: First submitted 2017-07-18; First posted 2017-07-26 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: [18F]DPA-714 PET scan — One PET scan using [18F]DPA-714 is done at M2 between two [123I]FP-CIT scan (DaTscan) done at M1 and M23.
  Neuropsychological assessment is done at M0, M18 and M24

SUMMARY:
Phase II, Open-labeled, Prospective, Multi-center study of assessing the link between microglial activation and dopaminergic denervation kinetics in the early stage of Parkinson disease, by using the imaging of [18F]DPA-714 a new ligand of Translocator Protein-18 kDa (TSPO) by Positron Emission Tomography (PET).

DETAILED DESCRIPTION:
The Parkinson's disease ( MP) is a frequent but heterogeneous neurodegenerative disease in term of clinical presentation(display) and evolutionary profile. The therapeutic coverage(care) of the patients would thus be personalized Such an approach remains still in its infancy in 2017. Better know the factors which determine the evolutionary clinical subcategories is a major question of the current researches on the Parkinson disease. Nigrostriaial inflammation is an interesting candidate. Microglia activation is closely associated with the degenerative process.

Development of the molecular imaging allows to study nigrostriatal inflammation in vivo in human by positron emission tomography (PET) by using the radiotracer of the protein of translocation of 18KDa ( TSPO), considered as a marker of microglia activation Some studies showed an increase of the inflammation in the striatum and in the substantia nigra, the sites of the dopaminergic degeneration (The lesional core of the Parkinson disease is the damage of the dopaminergic nigrostriatale way). However data remain rare and concern small number of patients. Some data are inconsistent because of problems of specificity of the ligands used and variation between populations of studied patients (duration of disease evolution).

In this study, investigators suggest studying by imaging TEP using a ligand new of the TSPO, [18F]DPA-714, microglial brain activation in the early stage of the Parkinson disease and determine wether it is predictive of speed of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a Parkinson's disease diagnosed according to the criteria UKPDSBB.
* Diagnosis done less than three years before the date the inclusion.
* Patient Age at diagnosis : between 40 and 65 years.
* Absence of clinical arguments for an associated neurovascular pathology.
* Written consent obtained.
* HAB polymorphism in the genotyping of TSPO gene.
* Brain MRI without following abnormalities: cortical or sub-cortical atrophy or hippocampal atrophy (Scheltens score ≥2), vascular encephalopathy (Fazekas score > 2, > 10 microbleed) or showing signs in favour of atypical parkinson syndrome.

Exclusion Criteria:

* Pregnant woman
* Minor
* Adult protected by the law
* Contraindication to PET-scan
* Contraindication to brain MRI
* History of inflammatory or dysimmune chronic disease
* History of psychiatric disease or drug addiction
* History of cognitive disorders (MMS<26)
* Hypersensibility to iodine derivates or one of these components
* Long-term Treatments which can interfere in neuroinflammation process
* Treatments / substances susceptible to interfere with the 18F-DPA-714
* TSPO gene Polymorphisms rs6971 corresponding to groups of affinity of low affinity (LAB=Low Affinity Binder) or moderated MAB = Mixed Affinity Binder)
* Modification of diagnosis of Parkinson disease during follow-up, in particular towards an atypical parkinson-like syndrome

Ages: 40 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2024-05-06 (Estimated); Study Completion 2024-05-06 (Estimated)

PRIMARY OUTCOMES:
Coefficient of correlation between level of microglial striatal activation and the And the dopaminergic denervation kinetics | 24 months
  Coefficient of correlation between the striatal microglial activation level measured by PET imaging [binding potential (BP) of 18F-DPA-714 in the striatum] and dopaminergic denervation kinetics obtained from two 123I-FP-CIT (DaTscan) scans

SECONDARY OUTCOMES:
Analyze the relationship between the level of microglial activation in the black substance at the early stage of MP and the dopaminergic denervation kinetics | 24 months
  Will be estimated by imaging PET with [18F]DPA-714
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic symptoms (motors) | baseline
  The equivalent dose of cumulative L-Dopa
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic symptoms (motors) | 18 months
  The equivalent dose of cumulative L-Dopa
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic symptoms (motors) | 24 months
  The equivalent dose of cumulative L-Dopa
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic symptoms (motors) | Baseline
  MDS-UPDRS scale (part III "OFF" - Part III "ON" and part II)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic symptoms (motors) | 18 Months
  MDS-UPDRS scale (part III "OFF" - Part III "ON" and part II)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic symptoms (motors) | 24 Months
  MDS-UPDRS scale (part III "OFF" - Part III "ON" and part II)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic symptoms (motors) | baseline
  MDS-UPDRS scale (part IV)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic symptoms (motors) | 18 months
  MDS-UPDRS scale (part IV)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic symptoms (motors) | 24 months
  MDS-UPDRS scale (part IV)
Evaluate the link between the level of striatal microglial activation at inclusion and:the severity of dopaminergic symptoms (non-motors) | baseline
  QUIP RS
Evaluate the link between the level of striatal microglial activation at inclusion and:the severity of dopaminergic symptoms (non-motors) | 18 months
  QUIP RS
Evaluate the link between the level of striatal microglial activation at inclusion and:the severity of dopaminergic symptoms (non-motors) | 24 months
  QUIP RS
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (motor) | baseline
  MDS-UPDRS scale (part III ON : 3.1 ; 3.2 ; 3.9 to 3.13)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (motor) | 18 months
  MDS-UPDRS scale (part III ON : 3.1 ; 3.2 ; 3.9 to 3.13)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (motor) | 24 months
  MDS-UPDRS scale (part III ON : 3.1 ; 3.2 ; 3.9 to 3.13)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (motor) | baseline
  MDS-UPDRS scale (part II : 2.13 and part III : 3.11)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (motor) | 18 months
  MDS-UPDRS scale (part II : 2.13 and part III : 3.11)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (motor) | 24 months
  MDS-UPDRS scale (part II : 2.13 and part III : 3.11)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | Baseline
  MDS-UPDRS scale (part I)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 months
  MDS-UPDRS scale (part I)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 months
  MDS-UPDRS scale (part I)
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | baseline
  NMS SCALE
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 months
  NMS SCALE
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 months
  NMS SCALE
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | baseline
  Scopa-Aut Score
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 months
  Scopa-Aut Score
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 months
  Scopa-Aut Score
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | Baseline
  Evaluation of constipation according to Rome III criteria
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 months
  Evaluation of constipation according to Rome III criteria
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 months
  Evaluation of constipation according to Rome III criteria
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | Baseline
  Detection of hypotension
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 months
  Detection of hypotension
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 months
  Detection of hypotension
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | Baseline
  Detection of paradoxical sleep disorder, according to the questionnaire for the detection of REM sleep disorders
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 months
  Detection of paradoxical sleep disorder, according to the questionnaire for the detection of REM sleep disorders
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 months
  Detection of paradoxical sleep disorder, according to the questionnaire for the detection of REM sleep disorders
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | Baseline
  Epworth's Sleepiness Scale
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 Months
  Epworth's Sleepiness Scale
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 Months
  Epworth's Sleepiness Scale
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | baseline
  UPSIT test
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 Months
  UPSIT test
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | Baseline
  MoCA score
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 Months
  MoCA score
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 Months
  MoCA score
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | Baseline
  MATTIS scale
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 Months
  MATTIS scale
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 Months
  MATTIS scale
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | Baseline
  Anxiety symptoms assessed using Beck's anxiety inventory
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 months
  Anxiety symptoms assessed using Beck's anxiety inventory
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 Months
  Anxiety symptoms assessed using Beck's anxiety inventory
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | Baseline
  Symptoms of depression assessed using the Beck Depression
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 18 Months
  Symptoms of depression assessed using the Beck Depression
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of symptoms considered mainly non-dopaminergic (non-motor) | 24 Months
  Symptoms of depression assessed using the Beck Depression
Evaluate the relation between the level of striatal microglial activation at inclusion and the severity of dopaminergic denervation at baseline (DaTscan initial) | Baseline
  Dopaminergic denervation at inclusion will be measured by the binding potential (BP) of ioflupane (123I-FP-CIT) by regions of interest in the caudate and putamen of the striatum
Evaluate the link between the level of microglial activation in the black substance and outcome 3 to outcome 57 | 24 Months
  MDS-UPDRS scale
Evaluate the link between the level of microglial activation in the black substance and outcome 3 to outcome 57 | 24 Months
  QUIP questionnaire
Evaluate the link between the level of microglial activation in the black substance and outcome 3 to outcome 57 | 24 Months
  NMS questionnaire
Evaluate the link between the level of microglial activation in the black substance and outcome 3 to outcome 57 | 24 Months
  Scopa-Aut Score
Evaluate the link between the level of microglial activation in the black substance and outcome 3 to outcome 57 | 24 Months
  Rome III criteria
Evaluate the link between the level of striatal microglial activation and the level of activation in other brain regions (black substance, bridge and cortex) | 24 months
  The level of cortical microglial activation measured by fixation of the radioligand 18F-DPA-714, on some volumes of interest in the brain
Assess the relationship between the level of microglial activation in the extra-striatal cortical (cortex and brain stem) regions and the presence of non-motor and axial motor symptoms. | baseline
  Neurologic Evaluation
Assess the relationship between the level of microglial activation in the extra-striatal cortical (cortex and brain stem) regions and the presence of non-motor and axial motor symptoms. | 18 months
  Neurologic Evaluation
Assess the relationship between the level of microglial activation in the extra-striatal cortical (cortex and brain stem) regions and the presence of non-motor and axial motor symptoms. | 24 months
  Neurologic Evaluation
Evaluate the link between the level of nigrostriatal microglial activation and the serum level of biological markers of inflammation | Baseline
  The serum levels of 13 cytokines will be analyzed
Evaluate the link between the level of nigrostriatal microglial activation and the serum level of biological markers of inflammation Evaluate the relationship between the level of nigrostriatal microglial activation | 18 months
  The serum levels of 13 cytokines will be analyzed
Evaluate the link between the level of nigrostriatal microglial activation and the serum level of biological markers of inflammation | 24 months
  The serum levels of 13 cytokines will be analyzed
Evaluate the relationship between the level of nigrostriatal microglial activation and the serum uric acid level at 0, 18 and 36 months | Baseline
  Measurement of serum uric acid
Evaluate the relationship between the level of nigrostriatal microglial activation and the serum uric acid level at 0, 18 and 36 months | 18 months
  Measurement of serum uric acid
Evaluate the relationship between the level of nigrostriatal microglial activation and the serum uric acid level at 0, 18 and 36 months | 24 months
  Measurement of serum uric acid

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Nantes, Nantes
  - Centre Eugène Marquis, Rennes
  - CHU de Rennes, Rennes
  - CHU de Tours, Tours